CLINICAL TRIAL: NCT00927173
Title: A Prospective Multicenter Double Blind Randomized Controlled Trial to Explore the Tolerability, Safety and Efficacy of the H-Coil Deep Transcranial Magnetic Stimulation (TMS) in Subjects With Major Depression Disorder (MDD)
Brief Title: Evaluation of the Brainsway Deep Transcranial Magnetic Stimulation (TMS) H-Coil in the Treatment of Major Depression Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brainsway (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTP-0001-00; IL-MOH-HTA-4860
Record Dates: First submitted 2009-06-23; First posted 2009-06-24 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2013-02

CONDITIONS: Major Depressive Disorder
Keywords: TMS; Transcranial Magnetic Stimulation; MDD; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham (Sham Comparator): Sham treatment
  Interventions: Device: Brainsway H-Coil Deep TMS System (Sham treatment)
- Active (Active Comparator): Active Deep Transcranial Magnetic Stimulation treatment
  Interventions: Device: Brainsway H-Coil Deep TMS System

INTERVENTIONS:
Device: Brainsway H-Coil Deep TMS System — Deep Transcranial Magnetic Stimulation (DTMS) is a new form of TMS which allows direct stimulation of deeper neuronal pathways than the standard TMS. The H-coil is a novel DTMS coil designed to allow deeper brain stimulation without a significant increase of electric fields induced in superficial cortical regions
  Arms: Active
Device: Brainsway H-Coil Deep TMS System (Sham treatment) — In the sham treatment,the electrical field induced by the sham coil cannot invoke any action potentials and if no action potentials are induced, then the electric field is insignificant and there is no treatment effect on the brain.
  Arms: Sham

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of deep brain rTMS, (Transcranial Magnetic Stimulation), a new experimental procedure using the H-Coil, in subjects with Major Depressive Disorder that have been previously unsuccessfully treated with antidepressant medications.

DETAILED DESCRIPTION:
This study is a multicenter, randomized double blind, sham controlled study to evaluate the safety and efficacy of H-coil deep transcranial magnetic stimulation (dTMS) as a treatment for patients with major depressive disorder who have been previously unsuccessfully treated with antidepressant medications. Studies of repetitive transcranial magnetic stimulation (rTMS), typically using a figure-8 coil, have shown that stimulating superficial brain regions can be beneficial in treating major depression. Differing from traditional figure-8 coil, the H-coil is designed to stimulate deep brain regions related to motivation, reward, and pleasure. Preliminary studies have been conducted and seem to indicate that through stimulating certain brain areas with the H-coil, dTMS may have an antidepressant effect. The study population will consist of patients with major depressive disorder who have failed adequate medication treatment or shown significant intolerance to medications. The study duration is 18 weeks, with a 2 week period of weaning the patient off medication, followed by 4 weeks of 5 daily treatments and 12 weeks of biweekly treatments. Mood and mental state will be carefully monitored through standard psychological scales and rating during the drug taper-down and throughout treatment.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients.
* Men and women 22-68 years of age.
* Primary DSM-IV diagnosis of Major Depression, single or recurrent episode.
* Current depressive episode is less than 5 years duration.
* The patient did not respond to at least one but not more than four antidepressant treatments in the current episode.
* Patients who have not completed antidepressant trials due to intolerance to therapy of 2 or more anti-depressant medications in the current episode.
* Satisfactory safety screening questionnaire for transcranial magnetic stimulation.
* Patients not suffering from hypo or hyper-thyroidism based on pre-study TSH level or medically stabilized.
* Patients able to tolerate psychotropic medication washout and no psychotropics during the treatment, other than benzodiazepine at equivalent daily dose of up to 3 mg lorazepam.

Exclusion Criteria:

* A history of schizophrenia, any psychotic disorder, PTSD, bipolar disorder, OCD, eating disorders (e.g., anorexia nervosa, bulimia) or substance abuse
* A history of panic disorder, social anxiety disorder or personality disorder (such as antisocial, schizotypal, histrionic, borderline, narcissistic) as assessed by the investigator to be primary, causing a higher degree of distress or impairment than MDD.
* A history of any significant medical disease (i.e., cardiovascular, gastrointestinal, etc.)
* A history of seizures, at risk for seizure (e.g., history of significant head trauma with loss of consciousness for greater than or equal to 5 minutes or familial or personal history of epilepsy) or have been diagnosed with a seizure disorder.
* Undergone rTMS treatment, Vagus Nerve Stimulation, or Deep Brain Stimulation.
* Received ECT within the last 3 months or failed to respond to ECT treatment.
* Individuals with a significant neurological disorder or insult including:

  * Any condition likely to be associated with increased intracranial pressure
  * Space occupying brain lesion
  * Any history of seizure EXCEPT those therapeutically induced by ECT
  * History of cerebrovascular accident
  * Transient ischemic attack within two years
  * Cerebral aneurysm
  * Dementia
  * Parkinson's disease
  * Huntington's chorea
  * Multiple sclerosis
* Individuals with hearing loss.
* Any intracranial implant such as aneurysm clips, shunts, stimulators, cochlear implants, or electrodes, or any other metal object within or near the head, excluding the mouth, that cannot be safely removed.
* A cardiac pacemaker, implanted medication pump, intracardiac line, or acute, unstable cardiac disease.
* Use of fluoxetine within 6 weeks of the randomization visit.
* Use of a Monoamine Oxidase Inhibitor (MAOI) within 2 weeks of the randomization visit.
* Present suicidal risk as assessed by the investigator.
* Implanted neurostimulators.
* History of abnormal MRI.
* If participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the rTMS trial.
* Clinically significant laboratory abnormality, in the opinion of the Investigator based on CBC and biochemistry.
* Women of childbearing potential and not using a medically accepted form of contraception when engaging in sexual intercourse.
* Women: if pregnant, planning on becoming pregnant, or currently nursing.

Ages: 22 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2009-09; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
HDRS-21 | 5 weeks

SECONDARY OUTCOMES:
Response rate | 5 weeks
Remission rates | 5 weeks
Quality of Life | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yechiel Levkovitz, M.D, Principal Investigator — Shalvat Mental Health Center; Abraham Zangen, Dr., Principal Investigator — Weizmann Institute of Science
Locations (22):
- United States (14):
  - University of California (UCLA), Los Angeles, California
  - UC Davis Center for Mind & Brain, Sacramento and Davis, California
  - Smart Brain and Health, Santa Monica, California
  - Advanced Mental Health Care Inc. - Juno Beach, Juno Beach, Florida
  - Advanced Mental Health Care Inc. - Royal Palm Beach, Royal Palm Beach, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - McLean Hospital - TMS Services, Belmont, Massachusetts
  - Greater Nashua Mental Health Center, Nashua, New Hampshire
  - Neuropharmacology Services, New York, New York
  - Columbia University / New York State Psychiatric Institute, New York, New York
  - Duke Medical Center Department of Psychiatry & Behavioral Sciences, Durham, North Carolina
  - Medical Uni. Of South Carolina (MUSC), Charleston, South Carolina
  - Senior Adults Specialty Research, Austin, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
- Center for Addiction and Mental Health (CAMH), Toronto, Ontario, Canada
- EPS Ville-Evrard, Neuilly-sur-Marne, France
- Germany (2):
  - Universitätsklinikum Bonn, Klinik und Poliklinik für Psychiatrie und Psychotherapie, Bonn
  - Klinik für Psychiatrie und Psychotherapie, Ludwig-Maximilians-Universität, Munich
- Israel (4):
  - Beer Yaacov Mental Health Center, Beer Yaacov
  - Shalvata Mental Health Center, Hod HaSharon
  - Hadasah Ein-Karem Medical Center, Jerusalem
  - Kfar Shaul Mental Health Center, Jerusalem